CLINICAL TRIAL: NCT01781832
Title: Evaluation of Pediatric Urinary Bladder Wall Thickening and Fibrosis Using Acoustic Radiation Force Impulse (ARFI)-Derived Shear Wave Velocities
Brief Title: Bladder ARFI (Acoustic Radiation Force Impulse) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ethan Smith, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00064416
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Bladder Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- (ARFI)-Derived Shear Wave Velocities (Experimental): This is an ultrasound-based new technique using Acoustic Radiation Force Impulse (ARFI). Shear Wave speeds are derived using ARFI.
  During ultrasound scanning a sound wave is sent towards tissue. The tissue's movement in response to the wave is measured in Shear Wave Velocity, which can estimate tissue stiffness. This technique may help detect bladder wall thickness and fibrosis (thickening) in the urinary bladder of pediatric patients.
  Interventions: Device: ARFI-Derived Shear Wave Velocities

INTERVENTIONS:
Device: ARFI-Derived Shear Wave Velocities — An ultrasound based scan uses ARFI, an acoustic radiation force impulse to estimate shear wave velocities during scanning of the urinary bladder. The research ultrasound scan lasts about 10 to 15 minutes.

SUMMARY:
Urinary bladder fibrosis (thickening and scarring) is fairly uncommon in children. Traditionally, the presence of urinary bladder fibrosis has been confirmed directly with bladder biopsy or using urodynamic testing. In this study we will use ultrasound scanning and ARFI (acoustic radiation force impulse) wave velocities to potentially identify any urinary bladder wall fibrosis.

DETAILED DESCRIPTION:
Urinary bladder fibrosis (thickening and scarring) is fairly uncommon in children. Traditionally, the presence of urinary bladder fibrosis has been confirmed directly with bladder biopsy or using urodynamic testing.

We will use ultrasound ARFI (acoustic radiation force impulse)-derived shear wave velocities to potentially identify the presence of urinary bladder wall fibrosis. We hypothesize that shear wave velocities found within the bladder wall will increase with increasing evidence of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or younger
2. Have an order for urodynamic testing from your doctor

Exclusion Criteria:

1. Adults
2. Unwilling to sign consent form

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Smith, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Having Urinary Testing: Subjects were pediatric patients scheduled to have a test on their bladder called CMG (cystometrogram). CMG is an invasive test that requires insertion of a catheter (tube) into the bladder.
  The patients agreed to have a research ultrasound (US) of their bladder. The US included a technique called elastography, which uses sound waves to measure the stiffness of tissue.
Period: Overall Study
Arm/Group | Subjects Having Urinary Testing
Started | 26
Completed | 25
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 26 subjects were included in this study.
Groups:
- (ARFI)-Derived Shear Wave Velocities: This is an new ultrasound-based technique using Acoustic Radiation Force Impulse (ARFI)-Derived Shear Wave Velocity Imaging. ARFI can be used to aid in detecting wall thickness and fibrosis in the urinary bladder of pediatric patients.
  ARFI-Derived Shear Wave Velocities: This technology uses ultrasound scanning with acoustic radiation force impulse-derived (called ARFI). This technique measures shear wave velocities to obtain and analyze images of the urinary bladder. The research ultrasound scan takes 10-15 minutes to complete.
Arm/Group | (ARFI)-Derived Shear Wave Velocities
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants] — The study location was a large tertiary pediatric hospital in the Midwest of the United States.
  Participants
    United States | 26
Age [Mean (Full Range); unit: years] | 4.6 [1 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Shear Wave Velocity, VTQ
Description: Shear wave velocity VTQ, or Virtual Touch Quantification is a "point" method for measuring a tissue's stiffness. A stiffness value is obtained from only the area in which a region of interest is placed.
Time Frame: Visit 0
Population: The subjects were pediatric patients already scheduled to have cystometrogram (CMG) testing for bladder abnormalities. CMG involves inserting a catheter into the urinary bladder.
  The ultrasound scans were investigated as an alternative way to determine bladder abnormalities. Ultrasound scanning is a non-invasive and painless procedure.
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- (ARFI)-Derived Shear Wave Velocities: This is an ultrasound-based new technique using Acoustic Radiation Force Impulse (ARFI)-Derived Shear Wave Velocity Imaging. This will aid in detecting bladder wall thickness and fibrosis in the urinary bladder of pediatric patients.
  ARFI-Derived Shear Wave Velocities: An ultrasound scan using acoustic radiation force impulse-derived shear wave velocities to obtain images of the urinary bladder. The research ultrasound scan l takes 15 minutes to complete. The shear wave velocity is a measure of the stiffness of the bladder wall.
Arm/Group | (ARFI)-Derived Shear Wave Velocities
Number analyzed (Participants) | 25
meters per second | 1.95 (0.63)

2. Primary Outcome: Shear Wave Velocity (VITQ)
Description: Shear Wave Velocity, VITQ, or Virtual Touch Tissue Imaging quantification is a color 2D method for measuring a tissues's stiffness. A color image (elastogram) of stiffness is acquired using this method. Then, one or more regions of interest can be placed in the area of interest on the elastogram. VITQ regions of interest are smaller than those used by VTQ.
Time Frame: Visit 0
Population: The subjects were pediatric patients already scheduled to have cystometrogram (CMG) testing for bladder abnormalities. CMG involves inserting a catheter into the bladder. The ultrasound scans may be an alternative way to determine bladder abnormalities. Ultrasound scanning is a non-invasive and painless procedure.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | (ARFI)-Derived Shear Wave Velocities
Number analyzed (Participants) | 25
meters per second | 2.37 (0.51)

ADVERSE EVENTS:
Time Frame: Subjects were observed for any adverse event at their sole visit.
Groups:
- (ARFI)-Derived Shear Wave Velocities: This is an ultrasound-based new technique using Acoustic Radiation Force Impulse (ARFI)-Derived Shear Wave Velocity Imaging. This will aid in detecting bladder wall thickness and fibrosis in the urinary bladder of pediatric patients.
  ARFI-Derived Shear Wave Velocities: An ultrasound based scan using acoustic radiation force impulse-derived shear wave velocities to obtain images of the urinary bladder. The research ultrasound scan will take approximately 10 to 15 minutes to complete.
Arm/Group | (ARFI)-Derived Shear Wave Velocities
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes